CLINICAL TRIAL: NCT00696995
Title: An Observational, Prospective Safety Study in Subjects With Type 2 Diabetes Mellitus Starting NovoMix® 30 (Biphasic Insulin Aspart) Treatment
Brief Title: An Observational Study of Type 2 Diabetes in Patients Starting on NovoMix® 30 Treatment
Acronym: Start
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-1917
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Venous blood samples drawn as part of routine clinical evaluation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Start dose and frequency as well as dose alterations to be determined by the physician according to normal clinical evaluation
  Other Names: NovoMix® 30

SUMMARY:
This study is conducted in Europe. The aim of this observational study is to evaluate the incidence of serious adverse drug reactions when initiating or switching to insulin therapy with NovoMix® 30 in subjects with type 2 diabetes under normal clinical practice conditions

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes
* Insulin-naive or previously treated by basal only insulin therapy

Exclusion Criteria:

* Patients who are unlikely to comply with the protocol
* Pregnancy or breastfeeding or intention of becoming pregnant

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The number of serious adverse drug reactions, including major hypoglycaemic events | at 26 weeks

SECONDARY OUTCOMES:
The number of all hypoglycaemic events | at 26 weeks
HbA1c | at 12 weeks and 26 weeks
Fasting plasma glucose at visits | at 12 weeks and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Lahti, Finland

REFERENCES:
- [Result] Makela JK, Schmuser C, Askonen K, Saukkonen T. Starting or switching to biphasic insulin aspart 30 (BIAsp 30) in type 2 diabetes: a multicenter, observational, primary care study conducted in Finland. Diabetes Res Clin Pract. 2012 Jan;95(1):10-8. doi: 10.1016/j.diabres.2011.06.006. Epub 2011 Nov 9. PMID 22078072
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com